CLINICAL TRIAL: NCT01777620
Title: A Study of Subject Satisfaction With BOTOX® Cosmetic Treatment in Facial Rhytides
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GMA-BTXC-12-001
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Facial Rhytides
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOTOX® (Active Comparator): BOTOX® (onabotulinumtoxinA) injected into the areas of glabellar lines and crow's feet lines on Day 1.
  Interventions: Biological: onabotulinumtoxinA
- Placebo (Placebo Comparator): Placebo (normal saline) injected into the areas of glabellar lines and crow's feet lines on Day 1.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: onabotulinumtoxinA — BOTOX® (onabotulinumtoxinA) injected into the areas of glabellar lines and crow's feet lines on Day 1.
  Other Names: botulinum toxin Type A; BOTOX®; BOTOX® Cosmetic
  Arms: BOTOX®
Drug: Normal Saline — Placebo (normal saline) injected into the areas of glabellar lines and crow's feet lines on Day 1.
  Arms: Placebo

SUMMARY:
This is a safety and efficacy study of BOTOX® in subjects with facial rhytides (glabellar lines and crow's feet lines).

ELIGIBILITY:
Inclusion Criteria:

* Glabellar lines and crow's feet lines
* No prior use of botulinum toxin therapy of any serotype for any reason

Exclusion Criteria:

* Previous facial cosmetic surgery, tissue grafting, or tissue augmentation with silicone or fat or other permanent fillers
* Planning a facial cosmetic procedure during the study period
* Diagnosis of myasthenia gravis, Eaton-Lambert Syndrome, and/or amyotrophic lateral sclerosis
* Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than study treatment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2013-05-29 (Actual); Study Completion 2013-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Toronto, Ontario, Canada

REFERENCES:
- [Background] Rivers JK, Bertucci V, McGillivray W, Muhn C, Rosen N, Solish N, Weichman BM, Wheeler S, Daniels SR, Gallagher CJ. Subject satisfaction with onabotulinumtoxinA treatment of glabellar and lateral canthal lines using a new patient-reported outcome measure. Dermatol Surg. 2015 Aug;41(8):950-9. doi: 10.1097/DSS.0000000000000424. PMID 26218728

RESULTS

PARTICIPANT FLOW:
Groups:
- BOTOX®: BOTOX® (onabotulinumtoxinA) 44U total dose injected into the areas of glabellar lines and crow's feet lines on Day 1.
Period: Overall Study
Arm/Group | BOTOX® | Placebo
Started | 63 | 62
Completed | 62 | 62
Not Completed | 1 | 0
Not completed — Subject Withdrawal | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the Per-Protocol population that included all randomized participants who received study treatment and had at least one post-baseline efficacy assessment and no major protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | BOTOX® | Placebo | Total
Number analyzed (Participants) | 60 | 57 | 117
Age, Customized [Number; unit: Participants]
  < 45 years | 25 | 24 | 49
  45 - 65 years | 35 | 33 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 50 | 98
  Male | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Satisfied With Treatment of Glabellar Lines Assessed Using the Facial Line Satisfaction Questionnaire (FLSQ)
Description: Participants assessed their overall satisfaction with their glabellar (frown) lines using the FLSQ 5-point scale where: -2=Very dissatisfied, -1=Mostly dissatisfied, 0=Neither dissatisfied nor satisfied, 1=Mostly satisfied and 2=Very satisfied. The percentage of participants with responses mostly or very satisfied is reported.
Time Frame: Day 60
Population: Per-Protocol population included all randomized participants who received study treatment and had at least one post-baseline efficacy assessment and no major protocol deviations.
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 81.7 | 0.0

2. Secondary Outcome: Percentage of Participants Satisfied With Treatment of Crow's Feet Lines (CFL) and Glabellar Lines Assessed Using the FLSQ
Description: Participants assessed their overall satisfaction with both their CFL and glabellar lines using the FLSQ 5-point scale where: -2=Very dissatisfied, -1=Mostly dissatisfied, 0=Neither dissatisfied nor satisfied, 1=Mostly satisfied and 2=Very satisfied. The percentage of participants mostly or very satisfied is reported.
Time Frame: Day 60
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 81.7 | 0.0

3. Secondary Outcome: Percentage of Participants Satisfied With Duration of Treatment of Glabellar Lines Assessed Using the FLSQ
Description: Participants assessed their overall satisfaction with duration of treatment of glabellar lines using the FLSQ 5-point scale where: -2=Very dissatisfied, -1=Mostly dissatisfied, 0=Neither dissatisfied nor satisfied, 1=Mostly satisfied and 2=Very satisfied. The percentage of participants with responses mostly or very satisfied is reported.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 65.0 | 0.0

4. Secondary Outcome: Percentage of Participants Where Treatment of Glabellar Lines Met Expectation Assessed Using the FLSQ
Description: Participants assessed whether treatment of their glabellar lines met expectation using the FLSQ 3-point scale where: 1=Worse than expected, 2=Met expectations and 3=Better than expected. The percentage of participants with responses Met expectations and Better than expected is reported.
Time Frame: Day 60
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 88.3 | 14.0

5. Secondary Outcome: Percentage of Participants Satisfied With Duration of Treatment of CFL and Glabellar Lines Assessed Using the FLSQ
Description: Participants assessed their overall satisfaction with duration of treatment of both CFL and glabellar lines using the FLSQ 5-point scale where: -2=Very dissatisfied, -1=Mostly dissatisfied, 0=Neither dissatisfied nor satisfied, 1=Mostly satisfied and 2=Very satisfied. The percentage of participants with responses mostly or very satisfied is reported.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 61.7 | 0.0

6. Secondary Outcome: Percentage of Participants Where Treatment of CFL and Glabellar Lines Met Expectation Assessed Using the FLSQ
Description: Participants assessed whether treatment of glabellar lines met expectations using the FLSQ 3-point scale where: 1=Worse than expected, 2=Met expectations and 3=Better than expected. The percentage of participants with responses Met expectations and Better than expected is reported.
Time Frame: Day 60
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 86.7 | 15.8

7. Secondary Outcome: Percentage of Participants Who Were Likely to Continue Treatment of Glabellar Lines Assessed Using the FLSQ
Description: Participants assessed how likely they were to continue treatment of glabellar Lines using the FLSQ 5-point scale where: 1=Not at all, 2=A little bit, 3=Moderately, 4=Quite a bit and 5=Extremely. The percentage of participants with responses Moderately, Quite a bit and Extremely is reported.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 78.3 | 36.8

8. Secondary Outcome: Percentage of Participants Who Were Likely to Continue Treatment of CFL and Glabellar Lines Assessed Using the FLSQ
Description: Participants assessed how likely they were to continue treatment of CFL and glabellar Lines using the FLSQ 5-point scale where: 1=Not at all, 2=A little bit, 3=Moderately, 4=Quite a bit and 5=Extremely. The percentage of participants with responses Moderately, Quite a bit and Extremely is reported.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 78.3 | 31.6

9. Secondary Outcome: Percentage of Participants With a Score of None or Mild in the Investigator's Assessment of the Severity of Glabellar Lines at Maximum Frown Assessed Using the FWS
Description: The Investigator assessed the severity of the patient's glabellar lines at maximum frown using the 4-point Facial Wrinkle Scale (FWS) where: 0=none, 1=mild, 2=moderate, and 3=severe. The percentage of participants with a score of none or mild is reported.
Time Frame: Day 30
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 83.3 | 1.8

10. Secondary Outcome: Percentage of Participants With at Least a 1-Grade Improvement in the Investigator's Assessment of the Severity of CFL at Maximum Smile Assessed Using the FWS
Description: The Investigator assessed the severity of the patient's CFL at maximum smile using the 4-point FWS where: 0=none, 1=mild, 2=moderate, and 3=severe. The percentage of participants with at least a 1-Grade improvement from Baseline is reported.
Time Frame: Baseline, Day 30
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | BOTOX® | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of participants | 86.7 | 8.8

ADVERSE EVENTS:
Arm/Group | BOTOX® | Placebo
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/62
Other Adverse Events (participants affected / at risk) | 6/63 | 4/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=63) | Placebo (N=62)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=63) | Placebo (N=62)
Headache (Nervous system disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No